CLINICAL TRIAL: NCT02428036
Title: A Phase I Study of Repeated Intratumoral Administration of TBI-1401(HF10), a Replication Competent HSV-1 Oncolytic Virus, in Patients With Solid Tumors With Superficial Lesions
Brief Title: A Study of TBI-1401(HF10) in Patients With Solid Tumors With Superficial Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBI1401-01
Record Dates: First submitted 2015-04-16; First posted 2015-04-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Solid Tumor
Keywords: TBI-1401(HF10); HF10; HSV-1; Oncolytic virus; Oncolytic virotherapy; Phase I; Melanoma; Intratumoral administration
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBI-1401(HF10) - Cohort 1 (Experimental): Oncolytic virotherapy, intratumoral administrations of TBI-1401(HF10)
  Interventions: Biological: TBI-1401(HF10)
- TBI-1401(HF10) - Cohort 2 (Experimental): Oncolytic virotherapy, intratumoral administrations of TBI-1401(HF10)
  Interventions: Biological: TBI-1401(HF10)

INTERVENTIONS:
Biological: TBI-1401(HF10) — Patients will receive intratumoral administrations of TBI-1401(HF10). The dose is 1 mL of 1x10^6 TCID50/mL.
  Arms: TBI-1401(HF10) - Cohort 1
Biological: TBI-1401(HF10) — Patients will receive intratumoral administrations of TBI-1401(HF10). The dose is 1 mL of 1x10^7 TCID50/mL.
  Arms: TBI-1401(HF10) - Cohort 2

SUMMARY:
The purpose of this study is to determine whether TBI-1401(HF10), a spontaneously attenuated mutant of Herpes Simplex Virus Type 1 (HSV-1), is safe and tolerable in the treatment of solid tumors with superficial lesions.

DETAILED DESCRIPTION:
This is an open label, non-randomized, dose escalation Phase I study evaluating the repeated intratumoral administrations of the TBI-1401(HF10), a spontaneously attenuated mutant of HSV-1, in patients with solid tumors with superficial lesions (e.g., malignant melanoma and squamous cell carcinoma of the skin).

The study will evaluate the safety and tolerability of repeated intratumoral administrations of TBI-1401(HF10) at dose levels of 1 x 10^6 TCID50/dose (cohort 1) and 1 x 10^7 TCID50/dose (cohort 2) in Japanese patients. Three patients will be enrolled in each cohort. Patients in the each cohort will receive a total of four intratumoral administrations in the same lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid tumors with superficial lesions.
* Patients must have unresectable and standard therapies-resistant solid tumors.
* Patients must be ≥ 20 years of age.
* Patients must have a life expectancy ≥ 12 weeks.
* Patients must have measurable non-visceral lesion(s) that are evaluable by the mWHO response criteria.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Patients must have adequate key organ function (bone marrow, heart, lung, liver, renal, etc), as defined as

  * Absolute neutrophil count ≥ 1,500/μL.
  * Platelet count ≥ 100,000/μL.
  * Total bilirubin levels ≤ 1.5 x upper limit of normal (ULN).
  * AST/ALT levels ≤ 2.5 x ULN, or ≤ 5 x ULN if liver metastases are present.
  * creatinine ≤ 1.5 x ULN.
  * creatinine clearance (calculated) ≥ 60 mL/min/1.73 m^2 for patients with creatinine > 1.5 x ULN.
* Patients must have passed 4 weeks after the completion of prior therapy [except bone metastasis therapy], or passed 8 weeks if immuno checkpoint inhibitor was treated.
* Patients must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patients with a history of significant tumor bleeding, or coagulation or bleeding disorders.
* Patients with Grade 2 adverse events Grade 2 or greater, except alopecia, resulting from anticancer agents administered more than 4 weeks prior to TBI-1401(HF10) administration.
* Patients receiving anti-herpes medication [except local treatment such as ointment].
* Patients receiving steroids or immunosuppressive agents [except inhaled steroid].
* Patients with clinically evident Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C virus (HCV) infection.
* Patients receiving anti-platelet medication.
* Patients receiving anti-coagulation medication.
* Patients with presence or medical history of central nervous system metastasis.
* Patients with Grade ≥ 2 pre-existing neurologic abnormalities (CTCAE version 4.0).
* Patients with severe cardiac disorder or abnormal cardiac rhythm.
* Patients with psychiatric disorder or drug dependency which affects informed consent.
* Pregnant or breastfeeding women; women or men, having normal reproductive potential, who disagree with the protection of pregnancy within the timeframe of the study.
* Patients received any other investigational products within 4 weeks, or within 8 weeks if immuno checkpoint inhibitor was treated.
* Patients would limit compliance with study requirements, as determined by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (CTCAE version 4.0). | up to Week 16
  Adverse events will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE version 4.0).

SECONDARY OUTCOMES:
Overall tumor response (modified World Health Organization response criteria) | at Week 12
  Overall tumor response will be evaluated by modified World Health Organization (mWHO) response criteria in the measurable target lesion(s) and unmeasurable/evaluable target lesion(s).
Levels of antibody to HSV-1 | up to Week 12
  Anti-HSV-1 antibodies will be assessed in serum.

OTHER OUTCOMES:
Change in cytokine profiles in serum | up to Week 12
  Evaluation of cytokine profiles in serum by immunoassay.
Change in antitumor T-cell reactivity in serum | up to Week 12
  Antitumor T-cell reactivity in serum will be evaluated by flow cytometry.
Change in regulatory T-cell (Treg) population in serum | up to Week 12
  Treg population in serum will be evaluated by flow cytometry.
Histopathological response with TBI-1401(HF10) administrated tumor | at Week 12
  Core biopsies will be performed to evaluate the histopathological response with TBI-1401(HF10) administrated tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Naoya Yamazaki, Principal Investigator — National Cancer Center Hospital
Locations (1):
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided